CLINICAL TRIAL: NCT06077032
Title: Chlorhexidine and Garlic Extract as Potential Topical Virucidal Therapeutic Agents of Non-Genital Warts: A Prospective, Randomized, Controlled, Blinded Clinical Trial
Brief Title: Chlorhexidine and Garlic Extract as Potential Topical Virucidal Therapeutic Agents of Non-Genital Warts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Nassar Abd El Hameed Ali, Assuit seed street, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: treatment of non genital warts
Record Dates: First submitted 2023-09-09; First posted 2023-10-11 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Non-Genital Warts
MeSH Terms: interventions — Solutions; Chlorhexidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- garlic extract (Experimental): Garlic will be collected from Medicinal Plant station, Pharmacognosy Department, Faculty of Pharmacy, Assiut University.
  The fresh garlic bulbs will be crushed. Extraction will be done using maceration method with Ethanol for 24 h at room temperature.
  Freeze-drying method will be used to remove solvent and give dry powder. Dry powder will be mixed with isopropyl alcohol in a ultrasonic bath to solve thoroughly.
  The soluble garlic extract will be added to a mixture of Polyethylene Glycol. The topical garlic formulation will be prepared for each time for two weeks-use and will be kept in dark glass containers in refrigerator till prescription.
  •Group 1: will apply Vaseline over the normal skin surrounding the lesion(s) then a cotton soaked with garlic extract (15%) solution will be applied under occlusion with a plastic tape for one hour and then washed by tap water daily for 6 weeks.
  Interventions: Drug: garlic extract (15%) solution
- chlorhexidine (Experimental): Chlorhexidine 4% (Laries, manufactured by: Smartec Egypt) will be diluted with equal amount of distilled water to obtain a concentration of 2%.
  •Group 2: will apply Vaseline over the normal skin surrounding the lesion(s) then a cotton soaked with topical chlorhexidine (2%) solution will be applied under occlusion with a plastic tape for one hour and then washed by tap water daily for 6 weeks.
  Interventions: Drug: topical chlorhexidine (2%) solution
- group3 (Placebo Comparator): •Group 3: (control) will use normal saline 0.9% as a placebo (they will be treated later on after completion of the study using any of the standard therapies for non-genital warts).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: garlic extract (15%) solution — •Group 1: will apply Vaseline over the normal skin surrounding the lesion(s) then a cotton soaked with garlic extract (15%) solution will be applied under occlusion with a plastic tape for one hour and then washed by tap water daily for 6 weeks.
  Arms: garlic extract
Drug: topical chlorhexidine (2%) solution — •Group 2: will apply Vaseline over the normal skin surrounding the lesion(s) then a cotton soaked with topical chlorhexidine (2%) solution will be applied under occlusion with a plastic tape for one hour and then washed by tap water daily for 6 weeks.
  Arms: chlorhexidine
Drug: Saline — •Group 3: (control) will use normal saline 0.9% as a placebo (they will be treated later on after completion of the study using any of the standard therapies for non-genital warts).
  Other Names: saline 0.9%
  Arms: group3

SUMMARY:
Aim(s) of the Research:

1. Evaluate the efficacy and safety of topical chlorhexidine (2%) solution vs garlic extract (15%) solution in treating non-genital warts.
2. Explore possible relation between therapeutic response with demographic/clinical data.
3. Identify patients satisfaction with each agent.

DETAILED DESCRIPTION:
Cutaneous warts or verruca are common, benign skin growths caused by human papilloma virus (HPV).

There are several therapeutic modalities for warts: include destructive agents (keratolytics, cryotherapy, curettage and cautery, laser, photodynamic therapy), antimitotic agents (podophyllin, bleomycin, retinoids), immune stimulants (topical sensitizers, cimetidine), and topical virucidal agents (formaldehyde, glutaraldehyde) Unfortunately, no single treatment is satisfactory for all patients. Chlorhexidine gluconate(CHX) is a gluconate salt with a broad-spectrum antiseptic action against Gram-Positive, Gram-negative bacteria, aerobes, facultative anaerobes, and fungi such action is mediated through increasing the permeability of the cell walls of microbes, causing their lysis.

Additionally, evidence indicates an in vitro effect against many viruses such as influenza A, parainfluenza, herpes virus 1, cytomegalovirus, hepatitis B, HIV and SARS-CoV-2.

It was hypothesized that the biophysiological mechanisms for the virucidal effect of CHX may be exerted through lysis of viral envelope, deterioration of nucleotide carbon chains, and inactivation and/or blocking of viral proteins.

Garlic (Allium sativum) is one of the most widely used medicinal plants with high therapeutic effects.

Clinical effectiveness of oral and topical garlic extract may be attributed to its antimicrobial, antioxidant, anti-inflammatory, anticancer and aging prevention effects.

However, the mechanisms of these actions are not clearly known. In vitro studies on garlic showed that garlic may enhance natural killer (NK) cells, which are an important part of the immune system in fighting cancers, viruses and certain bacteria.

Previous studies showed garlic extract was effective on complete resolution of cutaneous wart.

Chlorhexidine has not been used for treatment of warts in previous studies so we decided to explore its efficacy in treatment of warts.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the clinical diagnosis of common or plantar warts.

Exclusion Criteria:

* Pregnancy and lactation.
* Chronic systemic diseases such as chronic renal failure, hepatic insufficiency, and cardiovascular disorders.
* Patients with inflamed lesions
* Use of systemic or topical treatments during the last month before enrollment.
* Individuals with history of allergic reactions to garlic or chlorhexidine
* Patient with generalized dermatitis or allergic skin disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
●Evaluate the efficacy and safety of topical chlorhexidine (2%) solution vs garlic extract (15%) solution in treating non-genital warts | 6weeks up to 3 month
  will be evaluated by changing in the size (using ruler) and the number of lesions.
●Side effects (systemic of local) as burning, itching, erythema, pigmentary changes, ulceration, and scarring | 6weeks up to 3 month
  will be evaluated at each visit.

REFERENCES:
- [Background] Garcia-Oreja S, Alvaro-Afonso FJ, Sevillano-Fernandez D, Tardaguila-Garcia A, Lopez-Moral M, Lazaro-Martinez JL. A non-invasive method for diagnosing plantar warts caused by human papillomavirus (HPV). J Med Virol. 2022 Jun;94(6):2897-2901. doi: 10.1002/jmv.27514. Epub 2021 Dec 15. PMID 34890486
- [Background] Fernandez MDS, Guedes MIF, Langa GPJ, Rosing CK, Cavagni J, Muniz FWMG. Virucidal efficacy of chlorhexidine: a systematic review. Odontology. 2022 Apr;110(2):376-392. doi: 10.1007/s10266-021-00660-x. Epub 2021 Oct 12. PMID 34637092
- [Background] Brookes ZLS, Bescos R, Belfield LA, Ali K, Roberts A. Current uses of chlorhexidine for management of oral disease: a narrative review. J Dent. 2020 Dec;103:103497. doi: 10.1016/j.jdent.2020.103497. Epub 2020 Oct 17. PMID 33075450